CLINICAL TRIAL: NCT06055257
Title: Combination Therapy: Hyperbaric Oxygen and PENTOCLO for Treatment of Osteoradionecrosis of the Mandible, a Pilot Randomized Control Trial
Brief Title: Combination Therapy: Hyperbaric Oxygen and PENTOCLO for Treatment of Osteoradionecrosis of the Mandible
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: pending
Record Dates: First submitted 2023-09-06; First posted 2023-09-26 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Osteoradionecrosis; Osteoradionecrosis of Jaw; Osteoradionecrosis of the Mandible
Keywords: Osteoradionecrosis; ORN; PENtoxifylline, TOcopherol and CLOdronate; PENTOCLO; Hyperbaric Oxygen Therapy; HBOT; Head and Neck Cancer; Radiation Therapy
MeSH Terms: conditions — Osteoradionecrosis; Head and Neck Neoplasms | interventions — Pentoxifylline; Tocopherols; Clodronic Acid

STUDY DESIGN:
Intervention Model Description: Prospective, pilot, double blind, randomized (stratified to ORN stage), controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: One unblinded clinician will be required for management of side effects and dose adjustments of pentoxifylline and clodronate as required in the event of side effects or intolerance. However, all other participants including, patients, assessors, research team and data analysts will be blinded to group allocation. At standard follow-up examination, imaging and photographs will be taken and de-identified and then presented to a blinded oral and maxillofacial surgeon for EBA calculation and to a blinded radiologist for allocation of Notani classification grade.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Control) (Placebo Comparator): Standard of care treatment for ORN consisting of conservative measures (e.g. local irrigation, antiseptic mouthwash) and approximately 60 hyperbaric oxygen therapy (HBOT) treatments (90 minute exposures at 2.4 ATA each, scheduled Monday to Friday for 12 weeks - i.e., 5 treatments per week). At the conclusion of the study and at the discretion of the clinical team, patients randomized to the control group with residual disease may be considered for the mPENTOCLO protocol.
  Simultaneously, the 4-week mPENTOCLO "pre-treatment" phase will be started (as defined in the intervention section), followed by a sham/placebo mPENTOCLO treatment phase for a total of 12 months.
  Interventions: Drug: sham mPENTOCLO
- Group 2 (Intervention) (Experimental): Standard of care treatment as described for the control group (conservative measures and 60 HBOT treatments).
  Simultaneously, a comprehensive oral regimen (mPENTOCLO) will be started, including a 4-week "pre-treatment phase" followed by a "treatment phase" for a total of 12 months, as defined in the Intervention section.
  Interventions: Drug: modified PENTOCLO (mPENTOCLO)

INTERVENTIONS:
Drug: modified PENTOCLO (mPENTOCLO) — 4-week "pre-treatment" phase consisting of 2 g daily of Amoxicillin+Clavulanic acid 875/125 mg (1 g morning and night), 1 g ciprofloxacin (500 mg morning and night) and 50 mg Fluconazole daily (morning), taken orally by the patient.
  This is followed by an additional 11 months (12 months total) "treatment" phase consisting of 800 mg pentoxifylline (400 mg morning and night) and 800 IU tocopherol (400 IU morning and night) taken orally 5 days per week (Monday to Friday with no medications on Saturday and Sunday). If the patient deteriorates (i.e., worsening of ORN T 6 or 9-month follow-up) then clodronate 1600 mg once daily (Monday to Friday) for the rest of the study period will be added.
  Other Names: PENtoxyphylline, TOcopherol, and CLOdronate
  Arms: Group 2 (Intervention)
Drug: sham mPENTOCLO — 4-week "pre-treatment" phase consisting of 2 g daily of Amoxicillin+Clavulanic acid 875/125 mg (1 g morning and night), 1 g ciprofloxacin (500 mg morning and night) and 50 mg Fluconazole daily (morning), taken orally by the patient.
  This is followed by an additional 11 months (12 months total) of sham "treatment" phase (placebo).
  Other Names: Placebo
  Arms: Group 1 (Control)

SUMMARY:
Radiation is commonly used to treat cancer in the head and neck, however, this can lead to a serious complication called osteoradionecrosis (ORN), where there is necrotic (dead) open bone inside or outside of the mouth. This complication is difficult to treat, involves large healthcare costs, and can have devastating effects on quality of life.

Two common adjuncts used in treatment of ORN are hyperbaric oxygen therapy (HBOT), which may requires up to 60 treatments at a specialized clinic where patients are treated with high concentrations of oxygen using special chambers, and a less complex option called PENTOCLO which involves treating patients with several antibiotics followed by a combination of other oral medications taken for at least 1 year.

This pilot study will be guide the design of a definitive trial to examine if the combination of HBOT and a modified PENTOCLO protocol together is better than the current standard treatment of HBOT alone. Outcomes will include pain, side effects and the need for surgery in patients with ORN. Specifically, the results of this small, pilot study will help to inform the design of a future larger study.

DETAILED DESCRIPTION:
Osteoradionecrosis (ORN) of the mandible is a potentially devastating complication which can occur following radiation therapy for head and neck cancers. ORN is difficult to treat using standard methods, and is associated with high healthcare costs and potentially dire impacts on quality of life. In addition to conservative measures (e.g. antibiotics, local irrigation, oral care) and surgical management, there are two established adjuvant treatments for ORN: hyperbaric oxygen therapy (HBOT) and an oral regimen called PENTOCLO, which consists of pre-treatment with oral antibiotics followed by prolonged treatment with a combination of PENtoxifylline, TOcopherol (Vitamin E) and CLOdronate.

This will be the first study to investigate the potential benefits of combining HBOT and a modified PENTOCLO regimen for treatment of ORN. This study is a prospective, pilot, open label, outcome blinded, randomized controlled trial where participants with a confirmed diagnosis of mandibular ORN will be randomized (1:1 in blocks of 4, stratified by ORN stage) to receive either the standard HBOT treatment or HBOT plus a modified PENTOCLO regimen.

The primary objective of this pilot trial is to determine feasibility of a larger definitive trial by assessing recruitment, adherence to the interventional protocol, ability to achieve 12 months follow up, feasibility of completing outcome measures, and study costs (including research support and healthcare resources costs per patient). Clinical outcomes including improvement or worsening of ORN of the mandible after 12-month treatment will also be assessed.

Participants will be followed for 12 months from the start of treatment, with follow-ups at 4 weeks, 5/6 weeks, and 3, 6, 9, and 12 months to assess pain scores, ORN characteristics, quality of life and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mandibular ORN after completion of radiotherapy
* ORN will be defined as "an area of exposed devitalized irradiated bone (> 20 mm2)"; minor bone spicules (MBS) (< 20 mm2) in the absence of radiographic abnormality, will be considered clinically insignificant
* Has no contraindications for undergoing hyperbaric oxygen therapy as assessed by a Hyperbaric Physician, and is willing to commit the time to undergo 60 sessions
* Negative Human Chronic Gonadotropin (hCG) screening test at baseline (for female patients of reproductive age not practicing medically acceptable methods of birth control (e.g., hormonal contraceptives, implants, injectables, intrauterine device (IUD), intrauterine system (IUS), vasectomy and bilateral tubal ligation)
* Baseline in-date ECG (within 60 days prior to enrolment)
* Age ≥ 18

Exclusion Criteria:

* Inability to give informed consent
* Previous treatment for ORN (PENTOCLO, HBOT or surgery)
* Major surgical procedure planned (more extensive than sequestrectomy)
* Severe trismus and inability to obtain intraoral photographs
* Contraindications for HBOT: pneumothorax, bullous disease, uncontrolled hypertension, uncontrolled epilepsy, claustrophobia
* Contraindications to mPENTOCLO (inability to swallow medication; pregnancy or lactating; allergy to any study drug; currently on oral anticoagulants; hemorrhagic/coagulation disorder; Vitamin K deficiency; active unresolved cardiac disease; severe liver or kidney disease (CrCl<30 mL/min))
* Known QT prolongation as documented on an in-date ECG (within 60 days prior to enrolment) are excluded. Patients with the QTc prolongation associated with a correctable cause (e.g., electrolyte imbalance or drug-induced), and corrected QTc prior to enrolment into the study as documented on 12 lead ECG will be eligible for inclusion
* Patients requiring concurrent use of medications known to significantly prolong the QT interval with a high risk of clinical impact (e.g., erythromycin, cisapride, astemizole, pimozide or quinidine) are excluded unless safe discontinuation or substitution of these medications is feasible prior to initiation of the study
* Patients on medication with a potential but low risk of QTc prolongation (e.g., ondansetron, SSRIs) may be included if a post-initiation ECG conducted within 24-48 hours of starting ciprofloxacin or fluconazole confirms that there is no significant QTc prolongation
* History of cholestatic jaundice/hepatic dysfunction associated with amoxicillin-clavulanate
* Moderate to severe active liver disease (class B or C Pugh-Child Score) or active liver disease with significant acute elevation of LFT values
* History of myasthenia gravis
* Patients with a history of nontraumatic tendon disorders with severe functional impairment (i.e., significant swelling of the affected tendon, or partial tendon tear documented on clinical examination or imaging)
* Patients who have previously experienced peripheral neuropathy due to exposure to antibiotics
* Smokers, high alcohol intake (average of >2 standard drinks per day), sepsis, severe undernourishment and severe immunodeficiency conditions (e.g. HIV, autoimmune disease, immune-compromised)
* Persistent or recurrent cancer and active neoplastic pathology will be excluded
* Patients with documented Vitamin K deficiency
* Patients taking additional Vitamin E
* Patients with concomitant prescription of anti-resorptive or anti-angiogenic medications (e.g. risedronate, alendronate, aIbandronate, zoledronic acid, pamidronate, etidronate or prescription of denosusamab, etc.)
* Patients diagnosed with retinitis pigmentosa
* Patients diagnosed with clinically significant anemia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Recruitment and adherence to protocol (process) | Pilot study (including 12-month follow-up)
  Recruitment of two subjects per month on average over 12 months
Recruitment and adherence to protocol (process) | Pilot study (including 12-month follow-up)
  At least 70% of all eligible patients are recruited
Recruitment and adherence to protocol (process) | Pilot study (including 12-month follow-up)
  More than 80% of all recruited subjects complete 60 sessions of HBOT (20/24)
Recruitment and adherence to protocol (process) | Pilot study (including 12-month follow-up)
  More than 80% of patients in mPENTOCLO group complete mPENTOCLO protocol (10/12)
Recruitment and adherence to protocol (process) | Pilot study (including 12-month follow-up)
  80% 12-month follow-up rate (20/24)
Feasibility (resource) - Time | Pilot study (including 12-month follow-up)
  Investigators to keep logs of time required to perform study related work
Feasibility (resource) - Cost | Pilot study (including 12-month follow-up)
  Cost of study including research support and healthcare resource costs per patient

SECONDARY OUTCOMES:
Recovery from ORN at one-year follow-up | 12-month follow-up
  Proportion of patients reaching recovery within the study period in each group. "Recovery" will be defined as the absence of pain, pathologic fracture, and cutaneous fistula; exposed bone area (EBA) less than 20 mm2; and by evidence of stabilization or regression on radiographic findings (Notani classification score). Minor bone spicules of less than 20 mm2 that have no ongoing pain, and no radiographic abnormalities will be considered fully healed and not Notani grade 1.
Time required to achieve recovery in patients | Assessed at each scheduled follow-up (4 weeks, 5/6 weeks, and 3, 6, 9 and 12 months)
  Difference in time required to reach recovery in each group. "Recovery" will be defined as the absence of pain, pathologic fracture, and cutaneous fistula; exposed bone area (EBA) less than 20 mm2; and by evidence of stabilization or regression on radiographic findings (Notani classification score). Minor bone spicules of less than 20 mm2 that have no ongoing pain, and no radiographic abnormalities will be considered fully healed and not Notani grade 1.
Improvement and failure rates in patients treated in each group using an accepted clinical and radiographic scoring system: | Assessed at each scheduled follow-up (4 weeks, 5/6 weeks, and 3, 6, 9 and 12 months)
  Exposed bone area (EBA)
Improvement and failure rates in patients treated in each group using an accepted clinical and radiographic scoring system: | Assessed at each scheduled follow-up (4 weeks, 5/6 weeks, and 3, 6, 9 and 12 months)
  Notani Classification Score
  I ORN confined to dentoalveolar bone II ORN limited to dentoalveolar bone or mandible above the inferior dental canal, or both III ORN involving the mandible below the inferior dental canal, or pathological fracture, or skin fistula
Improvement and failure rates in patients treated in each group using an accepted clinical and radiographic scoring system: | Assessed at each scheduled follow-up (4 weeks, 5/6 weeks, and 3, 6, 9 and 12 months)
  Late Effects Normal Tissue Task Force-Subjective, Objective, Management and Analytic (LENT-SOMA) score
Complications that arise from treatment | Assessed at each scheduled follow-up (4 weeks, 5/6 weeks, and 3, 6, 9 and 12 months)
  Complications related to HBOT and/or mPENTOCLO, as defined in product monographs and study protocol.

OTHER OUTCOMES:
Quality of Life questionnaire | Assessed at each scheduled follow-up (4 weeks, 5/6 weeks, and 3, 6, 9 and 12 months)
  Assessed using EQ-5D-5L questionnaire
Xerostomia severity | Assessed at each scheduled follow-up (4 weeks, 5/6 weeks, and 3, 6, 9 and 12 months)
  Assessed using Xerostomia Inventory and/or Clinical Oral Dryness Score
Opioid usage | Assessed at each scheduled follow-up (4 weeks, 5/6 weeks, and 3, 6, 9 and 12 months)
  Medications and dosages (oral morphine equivalents) currently being taken by participants at each scheduled follow-up
ORN Pain | Assessed at each scheduled follow-up (4 weeks, 5/6 weeks, and 3, 6, 9 and 12 months)
  Assessed using Numerical Rating Scale (NRS) patient to rate their pain on scale of 0-10 where 0 is no pain and 10 is the worst pain imaginable

CONTACTS AND LOCATIONS:
Overall Officials: Ben Safa, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant-level data will be made available upon reasonable request to study PI following publication of full trial results.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: This is a pilot trial and full inferential analysis will not be conducted until completion of the full trial. As such, data will be available following publication of the primary results of the subsequent full trial.
Access Criteria: Data and supporting information will be made available following reasonable request directly to study PI.